CLINICAL TRIAL: NCT00712374
Title: Evaluation of the Public Health Impact and Cost Effectiveness of Seasonal Intermittent Preventive Treatment in Children in Senegal
Brief Title: Evaluation of the Public Health Impact of Seasonal Intermittent Preventive Treatment (IPT) in Children in Senegal
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Senegal: Ministere de la Sante (Unknown); Institut de Recherche pour le Developpement (Other Government); Cheikh Anta Diop University, Senegal (Other)
Responsible Party: Prof Oumar Gaye, Universite Cheikh Anta Diop
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PSP01; 40099
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Malaria
Keywords: Malaria; All causes mortality; Cost effectiveness
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Amodiaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Children 3 months to 10 years old will receive a treatment dose of SP+AQ on three occasions during the malaria transmission season, delivered by the local health post
  Interventions: Drug: sulfadoxine-pyrimethamine plus amodiaquine

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine plus amodiaquine — SP+AQ on three occasions during the malaria transmission season
  Intermittent Preventive Treatment with sulfadoxine-pyrimethamine plus amodiaquine

SUMMARY:
In areas of seasonal malaria transmission the burden of severe disease and mortality due to malaria is mainly among children under 5 years of age. Intermittent preventive treatment (IPT) with antimalarial drugs given to all children once a month during the transmission season is a promising new strategy for malaria prevention. Studies in Senegal, Ghana, Mali and The Gambia have shown this approach can be highly effective. In Senegal, seasonal IPT with sulfadoxine-pyrimethamine (SP) and one dose of artesunate resulted in a 90% reduction in incidence of clinical malaria in a recent trial in Senegal (Cisse et al., Lancet 2006). The purpose of the present project is to determine the public health impact and cost effectiveness of this intervention when it is delivered through the routine health service to communities in rural areas in Senegal. Demographic surveillance will be set up in the rural population of three districts (Mbour, Bambey and Fatick) which comprises approximately 540,000 people, including 100,000 children under 5 yrs, and is served by 54 health posts, as an expansion of the area covered by the existing DSS of Niakhar. Information about births, deaths and migrations, household characteristics such as socioeconomic status, and vaccination status of children and their use of bednets, will be recorded in 6-monthly rounds of all households. In selected areas, deaths among children under 10 years will be investigated using verbal autopsies. Over four years from September 2008 - November 2011, seasonal IPT (three monthly administrations of SP (sulfalene-pyrimethamine) plus amodiaquine during the transmission season each year to children 3-59 months of age) will be introduced gradually, in a step-wedge design, by 9 health posts in 2008, by an additional 18 posts in 2009, and another 18 in 2010 and 9 in 2011. At the end of each transmission season, a cross-sectional survey of 2400 children under 5 yrs of age, in which finger prick blood samples will be taken, will be used to estimate the prevalence of molecular markers of drug resistance to Plasmodium falciparum, the prevalence of anaemia and the nutritional status of children. Malaria incidence will be monitored by passive surveillance through health posts, health centres, and hospitals. Cost effectiveness will be assessed. Due to changes in the epidemiology of malaria in the study area, the upper age limit for inclusion was increased from 5 to 10 years old from September 2009.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-119 months at time of first administration of IPT in September
* Consent of mother or carer and the local community

Exclusion Criteria:

* History of allergy to SP or AQ
* Age < 3 months or >119 months at time of first administration of IPT in September

From 2009, the age for inclusion has been changed from 3-59 months to 3 months to 10 years of age.

Ages: 3 Months to 119 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100000 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-12 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
All-causes mortality | 2008-2010

SECONDARY OUTCOMES:
Incidence of malaria by passive case detection | 2008-2010

CONTACTS AND LOCATIONS:
Overall Officials: Oumar Gaye, PhD, Study Director — Universite CHeikh Anta Diop; Badara Cisse, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Cheikh Sokhna, PhD, Principal Investigator — IRD, Dakar; Oumar Faye, MD, Principal Investigator — Ministere de la Sante et de la Prevention; Paul Milligan, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine

REFERENCES:
- [Derived] Dieng S, Ba EH, Cisse B, Sallah K, Guindo A, Ouedraogo B, Piarroux M, Rebaudet S, Piarroux R, Landier J, Sokhna C, Gaudart J. Spatio-temporal variation of malaria hotspots in Central Senegal, 2008-2012. BMC Infect Dis. 2020 Jun 17;20(1):424. doi: 10.1186/s12879-020-05145-w. PMID 32552759
- [Derived] Cisse B, Ba EH, Sokhna C, NDiaye JL, Gomis JF, Dial Y, Pitt C, NDiaye M, Cairns M, Faye E, NDiaye M, Lo A, Tine R, Faye S, Faye B, Sy O, Konate L, Kouevijdin E, Flach C, Faye O, Trape JF, Sutherland C, Fall FB, Thior PM, Faye OK, Greenwood B, Gaye O, Milligan P. Effectiveness of Seasonal Malaria Chemoprevention in Children under Ten Years of Age in Senegal: A Stepped-Wedge Cluster-Randomised Trial. PLoS Med. 2016 Nov 22;13(11):e1002175. doi: 10.1371/journal.pmed.1002175. eCollection 2016 Nov. PMID 27875528
- [Derived] NDiaye JL, Cisse B, Ba EH, Gomis JF, Ndour CT, Molez JF, Fall FB, Sokhna C, Faye B, Kouevijdin E, Niane FK, Cairns M, Trape JF, Rogier C, Gaye O, Greenwood BM, Milligan PJ. Safety of Seasonal Malaria Chemoprevention (SMC) with Sulfadoxine-Pyrimethamine plus Amodiaquine when Delivered to Children under 10 Years of Age by District Health Services in Senegal: Results from a Stepped-Wedge Cluster Randomized Trial. PLoS One. 2016 Oct 20;11(10):e0162563. doi: 10.1371/journal.pone.0162563. eCollection 2016. PMID 27764102